CLINICAL TRIAL: NCT00039052
Title: An Open Label, Multiple-Dose, Sequential Dose-Escalation Study of NBI-3001 in Patients With Recurrent or Unresponsive Solid Tumors Known to Over-Express IL-4 Receptors
Brief Title: Intravenous Interleukin-4 PE38KDEL Cytotoxin in Treating Patients With Recurrent or Metastatic Kidney Cancer, Non-Small Cell Lung Cancer, or Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: NBI-3001-ST-0101; CDR0000069228 (Registry Identifier: PDQ (Physician Data Query)); UARIZ-HSC-01196; UCLA-0108085; NCI-V02-1692
Record Dates: First submitted 2002-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2003-03

CONDITIONS: Breast Cancer; Kidney Cancer; Lung Cancer
Keywords: stage IV breast cancer; recurrent breast cancer; recurrent non-small cell lung cancer; stage IV renal cell cancer; recurrent renal cell cancer; stage IV non-small cell lung cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Kidney Neoplasms; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Breast Neoplasms, Male | interventions — interleukin-4-Pseudomonas exotoxin

INTERVENTIONS:
Biological: interleukin-4 PE38KDEL cytotoxin

SUMMARY:
RATIONALE: Interleukin-4 PE38KDEL cytotoxin may be able to deliver cancer-killing substances directly to solid tumor cells.

PURPOSE: Phase I trial to study the effectiveness of intravenous interleukin-4 PE38KDEL cytotoxin in treating patients who have recurrent or metastatic kidney cancer, non-small cell lung cancer, or breast cancer that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of interleukin-4 PE38KDEL cytotoxin in patients with recurrent or unresponsive, metastatic renal cell, non-small cell lung, or breast cancer that overexpresses interleukin-4 receptors.
* Determine the qualitative and quantitative toxic effects of this drug, including the duration and intensity of these toxic effects, in these patients.
* Determine the pharmacokinetic behavior of this drug in these patients.
* Determine the antibody response (if any) in patients treated with this drug.
* Determine, in a preliminary manner, the antitumor activity of this drug in these patients.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive interleukin-4 PE38KDEL cytotoxin (NBI-3001) IV over 10 minutes once daily on days 1-5. Treatment repeats every 28 days in the absence of disease progression, unacceptable toxicity, or detection of neutralizing antibodies.

Cohorts of 3-6 patients receive escalating doses of NBI-3001 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

PROJECTED ACCRUAL: A maximum of 36 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent or unresponsive, metastatic renal cell, non-small cell lung, or breast cancer that has been treated previously with standard surgery, radiotherapy, chemotherapy, or immunotherapy or for which no available treatment options currently exist
* Confirmed overexpression of interleukin-4 receptors
* Measurable disease (lesions greater than 10 mm by CT scan) OR
* Evaluable disease
* No prior or concurrent clinically significant brain metastases
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Sex:

* Male or female

Menopausal status:

* Not specified

Performance status:

* Karnofsky 70-100%

Life expectancy:

* More than 12 weeks

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* Transaminases no greater than 1.5 times ULN
* Albumin at least 2.5 g/dL
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative
* No prior or concurrent hepatic disease (e.g., hepatitis or alcoholic liver disease)

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* See Surgery
* Electrocardiogram normal
* MUGA scan normal
* No congestive heart failure
* No cardiac arrhythmia requiring treatment
* No myocardial infarction
* No clinical evidence of coronary artery disease (unless there is a cardiac evaluation and evidence of adequate coronary function by a stress test or angiography)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 4 weeks before, during, and for at least 3 months after study
* No concurrent underlying medical condition that would preclude study or cannot be controlled
* No active infection

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* See Disease Characteristics

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy

Surgery:

* See Disease Characteristics
* At least 1 year since prior surgery or angioplasty for coronary artery disease

Other:

* At least 28 days since prior experimental drugs and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-01; Primary Completion 2003-05 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Pan, MD, PhD, Study Chair — Neurocrine Biosciences
Locations (2):
- United States (2):
  - Arizona Cancer Center, Tucson, Arizona
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California